CLINICAL TRIAL: NCT00664924
Title: Comparative In-patient, Non-intervention Study of the Remote Physiological Monitoring System (RPM™), a Non-invasive, Remote, Ambulatory Vital Signs Monitoring Device, Versus Standard Physiological Monitoring Devices by Simultaneous Monitoring of Heart Rate, ECG, SpO2, Blood Pressure, Body Temperature, and Respiration Rate in a 24 hr Monitoring Period (BRYTECH #BRY-C-01-06-RPM)
Brief Title: Comparative in Patient, Non-intervention Study of the Remote Physiological Monitoring System (RPM™) vs Standard Physiological Monitoring Devices
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: BryTech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BRY-C-01-06-RPM; OHREB #2006712-01H (Other: Ottawa Hospital Research Ethics Boards)
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Physiological Monitoring; Critically Ill
Keywords: ICU
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Remote Physiological Monitoring System (RPM™) is a wireless technology for physiological monitoring. The RPM™ is designed to capture, transmit and remotely monitor the vital signs of a patient or group of patients. The RPM™ allows the patient to carry an unobtrusive unit and sensor array, which is able to store and/or forward its data via existing communication networks. This data is archivable and can be made available to a monitoring station or stations. This approach obviates the need to provide new and expensive infrastructure to support the system since it is designed to 'piggy-back' on the existing network.

A major clinical advantage of the RPM™ and the principal reason why it may offer a benefit to patients, is that it provides continuous remote monitoring of vital signs, in contrast to the current situation for ward patients, where there is intermittent vital signs monitoring. This is a major advantage for patients and hospital staff, since there is increasing evidence that demonstrate early recognition and treatment of clinical events, e.g., shock, can save lives; the concurrent cost and labour saving is a further obvious benefit.

The RPM™ uses wireless technology to overcome the portability problems associated with conventional patient monitoring systems. The RPM™ consists of the following system components:

1. Physiological Monitoring Unit (PMU)
2. Data Aggregation Server (DAS)
3. Clinical Monitoring Position (CMP) To validate the RPM™ device for regulatory approval, BRYTECH will evaluate the RPM™ in a clinical setting, thereby ensuring that the system is trustworthy and acceptable to health professionals as a monitoring system in patients. The study proposes to evaluate the accuracy and reliability of the RPM™ compared to monitors commonly used in the medical practice under the standard conditions of medical practice The study also proposes to evaluate notification and alarm systems, the communications interface and non-interference with existing systems, devices, networks and procedures as well as the incremental nursing workload associated with the integration of the RPM™ in a clinical environment. The RPM™ and reference physiological monitoring devices will be compared for physiological monitoring capabilities in 40 patients.

DETAILED DESCRIPTION:
BRYTECH STUDY SUMMARY

The Remote Physiological Monitoring System (RPM™) is a wireless technology for physiological monitoring. The RPM™ is designed to capture, transmit and remotely monitor the vital signs of a patient or group of patients. The RPM™ allows the patient to carry an unobtrusive unit and sensor array, which is able to store and/or forward its data via existing communication networks. This data is archivable and can be made available to a monitoring station or stations. This approach obviates the need to provide new and expensive infrastructure to support the system since it is designed to 'piggy-back' on the existing network.

A major clinical advantage of the RPM™ and the principal reason why it may offer a benefit to patients, is that it provides continuous remote monitoring of vital signs, in contrast to the current situation for ward patients, where there is intermittent vital signs monitoring. This is a major advantage for patients and hospital staff, since there is increasing evidence that demonstrate early recognition and treatment of clinical events, e.g., shock, can save lives; the concurrent cost and labour saving is a further obvious benefit.

The RPM™ uses wireless technology to overcome the portability problems associated with conventional patient monitoring systems. The RPM™ uses off the shelf computer technology such as standard displays, as well as secure, wireless, 802.11 networking protocols and consists of the following system components:

1. Physiological Monitoring Unit (PMU)
2. Data Aggregation Server (DAS)
3. Clinical Monitoring Position (CMP)

To validate the RPM™ device for regulatory approval, BRYTECH will evaluate the RPM™ in a clinical setting, thereby ensuring that the system is trustworthy and acceptable to health professionals as a monitoring system in patients. The study proposes to evaluate the accuracy and reliability of the RPM™ compared to monitors commonly used in the medical practice under the standard conditions of medical practice; this study will therefore be a non-intervention study. The study also proposes to evaluate notification and alarm systems, the communications interface and non-interference with existing systems, devices, networks and procedures as well as the incremental nursing workload associated with the integration of the RPM™ in a clinical environment. The RPM™ and reference physiological monitoring devices will be compared for physiological monitoring capabilities in 40 patients from the following four (4) cohorts:

1. Cohort 1 (Exercise): patients who are scheduled to undergo a minimum of 20 minutes of exercise testing.
2. Cohort 2 (ICU): patients admitted to the Intensive Care Unit (ICU)
3. Cohort 3 (Post-op): patients in Post-Operative care
4. Cohort 4 (ER): patients admitted to the Emergency Room (e.g., high risk medical admissions) These cohorts are considered representative of a broad spectrum of the general patient population. Patients participating in the study will be assigned to one of these 4 cohorts, with a minimum of 10 patients assigned to Cohort 1 (Exercise) and a minimum of 5 patients in each of the other cohorts.

For the study, the RPM™ and reference monitoring devices will be time-stamped such that zero time will be readily evaluable and patients will be fitted with all necessary sensors for collection of vital signs, namely heart rate (HR), electrocardiogram (ECG), blood oxygen saturation levels (SpO2), non-invasive blood pressure (NIBP), body temperature (BT) and respiration rate (RR).

For Cohort 1 (Exercise) patients, comparative monitoring of vital signs will be done during exercise testing for a minimum of 20 minutes with additional monitoring performed pre- and post-exercise. There will be a minimum of 10 patients in this cohort. For patients in Cohorts 2, 3 and 4, comparative monitoring of vital signs will be performed during the period (24 - 72 hours) required to collect 12 Vital Sign Assessment Cycles (VSAC - defined in Section 5.2.2) per subject, with a minimum of 5 patients in each cohort and a total of 30 patients. The four cohorts of patients have been chosen to allow comparison of vital signs from the RPM™ and standard nursing measurement techniques over a broad range of physiologic data (e.g. rest and exercise) and patient populations (e.g. stable and critically ill).The primary objective for the study is to determine substantial equivalence of the RPM™ and the reference devices or standard practice measurements by comparing the agreement (accuracy) between paired output results for individual vital signs and the reliability of data collection over a 24 hour monitoring period. Timepoint matched paired data for all available timepoints will be collected from the RPM™ and the reference devices, excluding ambulatory data, for heart rate, ECG, SpO2, blood pressure, body temperature and respiration rate. Accuracy will be determined by assessing whether the paired values show significant agreement. Reliability will be determined by a comparison of cumulative totals for lost data points and error rates.

The study will be conducted according to Good Clinical Practice (GCP) guidelines with all patients required to sign an Informed Consent Form (ICF). This is a non-intervention study and patients tested will be subjected to use of the RPM™ as the only experimental procedure during the trial. Importantly, patients will not be exposed to any significant risks as a result of participating in this study.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent document must be read, signed, and dated by the patient (or legally authorized representative), the individual obtaining the consent, and a witness if appropriate, before conducting any study related procedures or examinations.
2. Patients will be ≥18 years of age or older, of any race and either sex. Women who are pregnant may participate in the study.
3. The RPM™ must not interfere with patient care.
4. Investigator or Study Staff must be able to clearly access the sites for attaching sensors.

Specific Inclusion Criteria for Cohort 1 (Exercise):

* Patients who are referred for Stage-I pre-operative exercise testing to assess fitness for surgery.
* Patients who have a history of a chronic respiratory or cardiac condition resulting in symptoms with exertion.

Specific Inclusion Criteria for Cohort 2 (ICU):

� Patients admitted to the ICU on life support whose hospital stay is expected to be more than 72 hours.

Specific Inclusion Criteria for Cohort 3 (Post-op):

* Patients undergoing surgery and post-operative recovery are expected to be more than 72 hours.
* A broad variety of patients with a history of coronary heart disease, congestive heart failure or chronic lung disease, and considered at high risk of cardiopulmonary complications; or patients who have undergone major thoracic surgery with a high risk of cardiopulmonary complications.

Specific Inclusion Criteria for Cohort 4 (ER):

� Patients who are admitted to a general medical ward from the ER whose hospital stay is expected to be more than 72 hours.

Exclusion Criteria:

1. Patients with a history of any medical condition which would preclude completion of the study, e.g., patients whose skin disorders or excessive weight interfere with the proper functioning of standard monitoring.
2. Patients with significant unstable disease that could compromise the study assessments and/or participation in the study.
3. The PI or the Medical Monitor may declare a patient ineligible for a valid medical reason or where the patient's condition or patient's actions may be inappropriate for inclusion in a study of this design.

Specific Exclusion Criteria for Cohort 1 (Exercise):

* Patients who would not tolerate a standard exercise test such as patients who have severe peripheral vascular disease, disabling arthritis or neurological condition;
* Patients who have had a significant change in symptoms since referral (e.g., unstable angina, recent myocardial infarction).

Specific Exclusion Criteria for Cohort 2 (ICU), 3, & 4:

* Patients who are severely agitated;
* Patients where increased monitoring may interfere with the provision of clinical care;
* Patients where the family or the attending team are not committed to providing all necessary aggressive supportive care;
* Patients who are considered brain dead;
* Patients where standard sensors are not capturing such as unstable patients with severe peripheral vascular disease where saturation probes do not function properly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1 (Exercise): patients who are scheduled to undergo a minimum of 20 minutes of exercise testing.
  Cohort 2 (ICU): patients admitted to the Intensive Care Unit (ICU) Cohort 3 (Post-op): patients in Post-Operative care Cohort 4 (ER): patients admitted to the Emergency Room (e.g., high risk medical admissions) These cohorts are considered representative of a broad spectrum of the general patient population. Patients participating in the study will be assigned to one of these 4 cohorts, with a minimum of 10 patients assigned to Cohort 1 (Exercise) and a minimum of 5 patients in each of the other cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
measurement and accurate transmission of data | June 2008

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Seely, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada